CLINICAL TRIAL: NCT04898322
Title: A Phase IIa Randomized, Double-blind, Parallel Group, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of Multiple Intravenous Injection of SY-005 in Sepsis Subjects
Brief Title: SY-005 （Recombinant Human Annexin A5）in Patients With Sepsis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SY005002
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2.5mg SY-005 (Experimental)
  Interventions: Drug: SY-005
- 5mg SY-005 (Experimental)
  Interventions: Drug: SY-005
- 10mg SY-005 (Experimental)
  Interventions: Drug: SY-005
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SY-005 — 2.5mg of SY-005 for each dose，doses to be given every 12 hours over a period of 5 days
  Arms: 2.5mg SY-005
Drug: SY-005 — 5mg of SY-005 for each dose，doses to be given every 12 hours over a period of 5 days
  Arms: 5mg SY-005
Drug: SY-005 — 10mg of SY-005 for each dose，doses to be given every 12 hours over a period of 5 days
  Arms: 10mg SY-005
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This Phase IIa Randomized, Double-blind, Parallel Group, Placebo-controlled, multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of Multiple Intravenous Injection of SY-005（recombinant human annexin A5） in Sepsis Subjects. 96 patients will be entered into the study and randomised in a 1:1:1:1 ratio to receive SY-005 2.5mg or SY-005 5mg or SY-005 10mg or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients are diagnosed with sepsis and receive study treatment within 48 hours
* Sepsis-related Organ Failure Assessment（SOFA）score range from 2 to 13
* The informed consent form signed by the patient or the patient's legally acceptable representative

Key Exclusion Criteria:

* Pregnant or breastfeeding women ; Women of childbearing potential (WOCBP) could not take effective method of contraception
* Moribund, and death is considered imminent within 24 hours or patient expected survival time is less than 6 months due to the underlying disease
* Absolute neutrophil count (ANC) <0.5 x 10^9/L
* New York Heart Association (NYHA) classification IV
* Patient with end-stage lung disease
* eGFR <60ml/min
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3.0 times the upper limit of normal (ULN)
* Immunosuppressed patients with following situations:

  1. Human immunodeficiency virus (HIV) infection
  2. Patients undergoing active radiation or chemotherapy treatment within the past 3 months
  3. Any organ or bone marrow transplant and related immunosuppressive therapy
  4. High dose steroids (eg, > 0.5 mg/kg prednisone or a steroid with equivalent activity, daily for a month) within 3 months before provision of written informed consent for the study
* Patients with high bleeding risk:

  1. Recent surgery <72 hours, or a planned surgical procedure in the next 24h
  2. Severe thrombocytopenia (< 30 x 10^9/L, before platelet transfusion)
  3. Recent trauma <72 hours
  4. History of gastrointestinal bleeding or intracranial hemorrhage in the past 6 weeks.
  5. Stroke or head injury in the past 3 months
  6. On-going therapeutic anticoagulants that could not be interrupted (except prophylactic heparin treatment that can be continued）
  7. Any history of Chronic liver disease with a Child score B or C
  8. Any condition at risk of bleeding, as appreciated by the physician in charge of the patient
* Severe anemia (hemoglobin <5.9 g/dL)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Parameters of SY-005 | From Day 0 to Day 28
  Number of patients with treatment-emergent adverse events over 28 days

SECONDARY OUTCOMES:
Change From Baseline in Sequential Organ Failure Assessment (SOFA) Score at Day 1, Day3, Day5, Day7 | Baseline, Day 1, Day3, Day5, Day7
Vasopressin Free Days From Day 0 to Day 28 | From Day 0 to Day 28
Assessment of ICU-Free Days From Day 0 to Day 28 | From Day 0 to Day 28
Ventilator-Free Days From Day 0 to Day 28 | From Day 0 to Day 28
7-Day and 28-Day Mortality | Over 7/28 Days Following First Dose
Change From Baseline in IL-1β at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in IL-6 at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Procalcitonin at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Prothrombin Time at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Thrombin Time at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Activated Partial Thromboplastin Time at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Fibrinogen at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Chemokine(C-C motif) Ligand 2 at Day 3，Day5 | Baseline, Day 3，Day5
Change From Baseline in Anti-drug Antibodies at Day7，Day14，Day28 | Baseline, Day7，Day14，Day28

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital，Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided